CLINICAL TRIAL: NCT06857149
Title: Effect of Cırcadıan Feedıng on Growth Parameters of Preterm Newborn
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayse Sonay Turkmen, Prof.Dr (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Ayse Sonay Turkmen, Prof.Dr, Assoc. Prof., Karamanoğlu Mehmetbey University
Organization: Karamanoğlu Mehmetbey University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Circadian Feeding
Record Dates: First submitted 2025-02-10; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Milk Expression, Breast; Nutrition
Keywords: Circadian feeding; Growth; Human milk; newborn
MeSH Terms: conditions — Breast Milk Expression | interventions — Milk, Human; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Circadian Rhythm Group (Experimental): In accordance with the physiology of breastfeeding, mothers will be asked to milk and deliver their milk to the ICU once every 3 hours. The mother will be asked to completely empty her breast with a milking machine. Before milking, the mother will wash her hands, and the parts of the milking machine that come into contact with the milk will also be boiled and disinfected after it is provided to be used. The mother will put the milk she has milked into a milking bag and deliver it to the researcher by writing the date and time on it. Feeding will be initiated by the neonatal specialist with the determination that the newborn is stable. During the period when mothers' babies are in the neonatal intensive care unit, the feeding of the babies in the circadian rhythm group will be carried out taking into account the date and day/night practice.
  The milk that the mother expresses at night will be given to her baby at night, and the milk that she expresses during the day will be used for day
  Interventions: Other: Human milk
- Experimental:Control Group (Active Comparator): The application in the control group is similar to the application in the cycadian rhythm group (mother's milking technique, collection method, storage and appropriate transportation, etc.) instead of the "milk expressed first is given first" condition used in routine practice, without taking into account the day and night characteristics of the expressed breast milk. will be brought. The routine practice of the clinic will continue. In line with the practice of the Turkish Neonatology Association (2018) and the clinic, the information of babies given breast milk fortifiers in the expressed breast milk of enterally fed babies will be recorded. In order to ensure that the data is collected safely and to facilitate monitoring, it will be recorded in the "Breastfeeding Follow-up Form", as in every feeding intervention group. The monitoring of babies is the same as in the circadian rhythm group. For the first month, the baby's weight and height will be measured and recorded twice a week.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Human milk — In accordance with the physiology of breastfeeding, mothers will be asked to milk and deliver their milk to the ICU once every 3 hours. The mother will be asked to completely empty her breast with a milking machine. Before milking, the mother will wash her hands, and the parts of the milking machine that come into contact with the milk will also be boiled and disinfected after it is provided to be used. The mother will put the milk she has milked into a milking bag and deliver it to the researcher by writing the date and time on it. Feeding will be initiated by the neonatal specialist with the determination that the newborn is stable. During the period when mothers' babies are in the neonatal intensive care unit, the feeding of the babies in the circadian rhythm group will be carried out taking into account the date and day/night practice.
  The milk that the mother expresses at night will be given to her baby at night, and the milk that she expresses during the day will be used for dayt
  Arms: Experimental:Circadian Rhythm Group
Other: Control Group — The application in the control group is similar to the application in the cycadian rhythm group (mother's milking technique, collection method, storage and appropriate transportation, etc.) instead of the "milk expressed first is given first" condition used in routine practice, without taking into account the day and night characteristics of the expressed breast milk. will be brought. The routine practice of the clinic will continue. In line with the practice of the Turkish Neonatology Association (2018) and the clinic, the information of babies given breast milk fortifiers in the expressed breast milk of enterally fed babies will be recorded. In order to ensure that the data is collected safely and to facilitate monitoring, it will be recorded in the "Breastfeeding Follow-up Form", as in every feeding intervention group. The monitoring of babies is the same as in the circadian rhythm group. For the first month, the baby's weight and height will be measured and recorded twice a week.
  Arms: Experimental:Control Group

SUMMARY:
This study was planned as a randomized controlled experimental study to determine the effect of circadian feeding on the growth parameters of preterm newborns. The data of the study were collected from patients aged 32-34 in the Neonatal Intensive Care Unit (NICU) of Selçuk University Faculty of Medicine. It will consist of premature babies and mothers born during the first week of gestation. The sample size was planned to include 48 preterm newborns and their mothers. Mother-Preterm Introductory Information Form, Breast Milk Feeding Follow-up Form, Breast Milk Content Parameters Follow-up Form, Newborn Baby Follow-up Form, Baby scale and height meter will be used in data collection. Data will be used with SPSS 21.0 package program and Kolmogorov-Smirnov (K-S) test for normality. Chi square, independent sample t-test, paired simple t-test, Wilcoxon tests and analysis of variance in repeated measurements will be used in the analysis of the data.

The research was conducted in the following order. All permissions were obtained for data collection. Individual characteristics were obtained from family members and recorded in the questionnaire. Newborns in the study or control group were randomly determined according to the day of admission.

For the newborns in the study group, the milk expressed by the mother at night will be given to the baby at night, and the milk expressed during the day will be given to the baby for daytime feeding. During this one-month period, the baby's weight and height will be measured and recorded twice a week.

For the newborns in the control group, the condition of "expressed milk is given first", which is used in routine practice, will be fulfilled, regardless of the day and night characteristics of the expressed breast milk. During this one-month period, the baby's weight and height will be measured and recorded twice a week.

Measurements of all newborns were made at the same time of the day.

DETAILED DESCRIPTION:
Ethical and institutional permissions were obtained before starting to collect the data. Written consent will be obtained from all parents via a voluntary consent form. Newborns will be randomly selected into 2 groups.

Control Group: The intervention in the control group will be implemented without taking into account the day and night characteristics of expressed breast milk, fulfilling the condition of "first expressed milk is given first" used in routine practice.

Circadian rhythm group: It will consist of infants fed with cycadian rhythm with the condition of "milk expressed in the morning is given in the morning".

Hypotheses of the Study H0: Breastfeeding according to the circadian rhythm in preterm newborns has no effect on the baby's weight and height levels.

H1: Feeding preterm newborns with breast milk according to the circadian rhythm has an effect on the weight gain of the babies.

H2: Feeding preterm newborns with breast milk according to the circadian rhythm has an effect on the height of the babies.

Research Type: a randomized controlled experimental study Research Variables Independent variables: Delivery of expressed breast milk according to circadian rhythm Dependent variable: Baby's weight, height Control variables; Descriptive characteristics of mothers and babies The population of the study was 32-34 patients in the Neonatal Intensive Care Unit (NICU) of Selçuk University Faculty of Medicine. It will consist of premature babies and mothers born during the first week of gestation. The mothers to be included in the study will be divided into two groups: circadian rhythm and control groups. The sample size was G Power 3.1.1, using weight gain as a criterion in line with the literature. program, with a power of 95% and a significance level of 0.05, a total of 44 were calculated, including 22 circadian rhythms and 22 controls. Since it was thought that there might be a loss of cases, it was planned to increase the number of cases by 10% and include 24 total of 48 preterm newborns and their mothers in each group.

Randomized controlled experimental studies, the permutation method is used to ensure that the number of cases in each group is balanced or equal, as well as to show a similar distribution in terms of some characteristics. In this method, block sets; are produced for each combination of identified prognostic factors. Providing equal distribution among the layers in terms of some features also increases the reliability of the study. Stratification was applied according to the gender of the baby. The groups represented by the letters were determined by the lottery method at the beginning of the data collection process. Blinding Single (participant) blinding was used in the study.

Inclusion Criteria;

* The mother is healthy (without a history of preeclampsia, hypertension, diabetes, hepatitis B or C, HIV, tuberculosis, mastitis or oncological disease)
* The mother's age is 32-34. Having given birth between weeks of gestation and staying in a hospital hotel
* The postnatal age of the newborn is 7 days or more
* Babies fed by gavage and oral methods *In order for the preterm baby to be fed effectively and safely orally, it is necessary for the preterm baby to be able to coordinate sucking-swallowing as well as breathing. Gavage feeding is a priority in babies who achieve this coordination. In babies who are able to coordinate sucking, swallowing and breathing, oral feeding will be started after an assessment of readiness for oral feeding will be made.

Exclusion Criteria;

* The mother does not follow a special diet
* Mother is not a vegetarian
* Mother's non-smoking
* The mother must have a body mass index within normal limits (BMI = 18.50-24.99)
* The baby is lying in the neonatal intensive care unit,
* The mother's inability to breastfeed her baby and feeding her own milk by regularly milking it every three hours
* Fully enteral fed babies
* Milking the mother's milk with a milking machine
* The baby does not have a health problem that will require surgical treatment
* Breastfeeding of the mother's baby after discharge
* 10 Of the birth percentile curves according to the gestational week of the baby.-90. among the percentile (those with a normal birth weight according to gestational age: Appropriate for Gestational Age -AGA) Dec.

Exclusion Criteria;

* According to the intrauterine growth curve, the baby's birth weight is low
* Feeding the baby with mama
* Total parenteral fed babies
* Discontinuation of mother's milk during the study process
* The mother's medication (antibiotics, etc.) to receive the treatment
* Those who have a small birth weight according to the gestational Age of the baby (Small for Gestational Age - SGA) and those who have a large birth weight according to the gestational age (Large for Gestational Age -LGA) Criteria for Exclusion from the Study;
* During the data collection process, the mother's medication (antibiotics, etc.) to receive the treatment
* Your mother does not want to continue working
* Early start of additional food by the mother October Data Sources and Data Collection Method Data Collection Tools The "Mother-Preterm Introductory Information Form", "Breast Milk Feeding Tracking Form", "Breast Milk Content Parameters Tracking Form" and "Baby Tracking Form", which contains the sociodemographic characteristics of the mother and the characteristic features of the babies, with a tracking table, will be used.

Collection of Data:

Before Application It was planned within the scope of the scientific outputs of the TUBITAK 1001 Project dated 15.10.2023 and numbered 123S615 and the permits of the ethics committee and the institution were obtained. Study Clinical Trials.gov 'a' will be recorded. During the data collection, mothers of babies admitted to the neonatal intensive care unit of the hospital where the study was conducted after childbirth who meet the criteria for inclusion in the study will be informed about the purpose of the study, the confidentiality of the answers, where and how the data will be stored. The mothers' questions about the subject will be answered. Mothers who volunteer to participate in the study will be asked to fill out the 'Informed Consent Form' and their written consent will be obtained. Mothers who volunteer to participate in the study will be randomly assigned to circadian rhythm and control groups. The "Mother-Preterm Introductory Information Form" will be applied, in which information about mothers in both groups (age, income status, pregnancy history, etc.) and the baby (weight, height, gestation week, etc.) is asked. The filling time of the form is about 10 minutes and the form will be filled in with a face-to-face interview. All mothers included in the scope of the research will be provided with information about the conditions of milking, storage and transportation with an electric pump. Mothers will be supported by researchers and the first milking process will be performed by showing. The brochure was sent to 6 specialists in the field of child health and diseases. In accordance with the expert opinions, it was determined that the content was appropriate.

Order of Application The subsequent data collection stages for each group will be as follows. Circadian Rhythm Group: In accordance with the physiology of breastfeeding, mothers will be asked to milk and deliver their milk to the ICU once every 3 hours. The mother will be asked to completely empty her breast with a milking machine. Before milking, the mother will wash her hands, and the parts of the milking machine that come into contact with the milk will also be boiled and disinfected after it is provided to be used. The mother will put the milk she has milked into a milking bag and deliver it to the researcher by writing the date and time on it. Feeding will be initiated by the neonatal specialist with the determination that the newborn is stable. During the period when mothers' babies are in the neonatal intensive care unit, the feeding of the babies in the circadian rhythm group will be carried out taking into account the date and day/night practice.

The milk that the mother expresses at night will be given to her baby at night, and the milk that she expresses during the day will be used for daytime feeding. Breast milk will be given according to both the date and the concept of milk expressed day and night. According to the routine practice of the clinic, babies weighing less than 1250 grams are fed every 2 hours, and babies weighing more than 1250 grams are fed every 3 hours. The amount of fluid that the baby should receive daily is calculated according to the baby's weight and divided according to the feeding frequency (every 2 hours: 12 times; every 3 hours: 8 times) to calculate the amount of breast milk the baby should receive. the clinic, the information of babies given breast milk fortifiers in the expressed breast milk of enterally fed babies will be recorded. According to the clinic's practice, when the daily amount of fluid the baby needs reaches 120ml/kg/day; One (1) scoop of breast milk fortifier is added to 50 ml of breast milk for the first 3 days, and one (1) scoop to 25 ml of breast milk after the 3rd day. The mothers' milk 7 days after birth (transitional milk) will be used as the first analysis milk. Then, the milk expressed by the mother will be collected every 6 hours. After the milk delivered by the mother to the unit is mixed with a disposable plastic spoon, 5-10 ml will be reserved for necessary analysis. The separated milk will be evaluated and recorded in terms of fat, carbohydrates, protein, vitamins, melatonin and trace elements. The mother's milk will be analyzed once a week at 6-hour intervals for an average of 4 weeks (approximately 16 times in total). The reason why breast milk is collected once a week at 6-hour intervals (4 times a week) for 1 month is to detect changes during the day and to determine the long-term effect of these changes on growth. Breast milk taken from mothers will be blinded and delivered to a researcher specialized in analytical chemistry. Parameter values obtained after breast milk analysis will be recorded in the "Breast Milk Content Parameters Tracking Form". The baby's growth monitoring will be done in a suitable room in the NICU. The baby's weight and height will be monitored as growth parameters. Groups will be recorded in the "Baby Monitoring Form" in terms of weight change. During this period, the baby's weight and height will be measured and recorded twice a week. During the measurements, the baby's safety will be taken into consideration and all precautions will be taken against falls or dangers.

Control Group: The application in the control group is similar to the application in the cycadian rhythm group (mother's milking technique, collection method, storage and appropriate transportation, etc.) instead of the "milk expressed first is given first" condition used in routine practice, without taking into account the day and night characteristics of the expressed breast milk. will be brought. The routine practice of the clinic will continue. the clinic, the information of babies given breast milk fortifiers in the expressed breast milk of enterally fed babies will be recorded. In order to ensure that the data is collected safely and to facilitate monitoring, it will be recorded in the "Breastfeeding Follow-up Form", as in every feeding intervention group. The monitoring of babies is the same as in the circadian rhythm group. For the first month, the baby's weight and height will be measured and recorded twice a week.

After the application In the circadian rhythm and control groups, the recording process will be performed after ensuring the safety of the baby after each application. Planning will be made for the next meeting and goodbye will be said with the family.

Statistical analyses will be performed using the SPSS package program, version 21.0 (IBM SPSS Statistics). Kolmogorov-Smirnov (K-S) test will be used for normality. Chi-square, independent sample t-test, paired simple t-test, Wilcoxon tests and variance analysis for repeated measurements will be used in the analysis of the data. The results will be evaluated within the 95% confidence December.

ELIGIBILITY:
Inclusion Criteria:

* -The mother is healthy (without a history of preeclampsia, hypertension, diabetes, hepatitis B or C, HIV, tuberculosis, mastitis or oncological disease)
* The mother's age is 32-34. Having given birth between weeks of gestation and staying in a hospital hotel
* The postnatal age of the newborn is 7 days or more
* Babies fed by gavage and oral methods *In order for the preterm baby to be fed effectively and safely orally, it is necessary for the preterm baby to be able to coordinate sucking-swallowing as well as breathing (Tian et al. 2015). Gavage feeding is a priority in babies who achieve this coordination (TND, 2018). In babies who are able to coordinate sucking, swallowing and breathing, oral feeding will be started after an assessment of readiness for oral feeding will be made.

The Sampling Inclusion Criteria of the Study;

* The mother does not follow a special diet
* Mother is not a vegetarian
* Mother's non-smoking
* The mother must have a body mass index within normal limits (BMI = 18.50-24.99) (WHO, 2022b)
* The baby is lying in the neonatal intensive care unit,
* The mother's inability to breastfeed her baby and feeding her own milk by regularly milking it every three hours
* Fully enteral fed babies
* Milking the mother's milk with a milking machine
* The baby does not have a health problem that will require surgical treatment
* Breastfeeding of the mother's baby after discharge
* 10 Of the birth percentile curves according to the gestational week of the baby.-90. among the percentile (those with a normal birth weight according to gestational age: Appropriate for Gestational Age -AGA) Dec.

Exclusion Criteria:

* According to the intrauterine growth curve, the baby's birth weight is low
* Feeding the baby with mama
* Total parenteral fed babies
* Discontinuation of mother's milk during the study process
* The mother's medication (antibiotics, etc.) to receive the treatment
* Those who have a small birth weight according to the gestational Age of the baby (Small for Gestational Age - SGA) and those who have a large birth weight according to the gestational age (Large for Gestational Age -LGA)

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — preterm newborns
Enrollment: 48 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
height length | Once a week for 4 weeks
  the height length of the newborn will be measured (height in centimeters)
weight | Once a week for 4 weeks
  weight of the newborn will be measured (weight in kilograms).

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe S Türkmen, Principal Investigator — Karamanoğlu Mehmetbey University
Locations (1):
- Karamanoğlu Mehmetbey University, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No